CLINICAL TRIAL: NCT06184412
Title: Periodontal Status Assessment, Molecular Mechanisms Underlying Inflammatory Response, and Endothelial Dysfunction Evaluation in Patients With Polycystic Ovary Syndrome
Brief Title: Periodontal Status and Endothelial Dysfunction in Patients With Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Milagros Rocha Barajas, Senior Postdoctoral Researcher, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Other Study IDs: PI19/00437B
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Periodontal Diseases
Keywords: inflammation; atherosclerosis; gingivitis; oxidative stress
MeSH Terms: conditions — Periodontal Diseases; Inflammation; Atherosclerosis; Gingivitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group without periodontal disease: Women without periodontal disease neither PCOS
- PCOS group with or without periodontal disease: Women with PCOS with or without periodontal disease

SUMMARY:
Emerging research indicates a link between polycystic ovary syndrome (PCOS) and periodontal diseases, revealing the intricate relationship between oral health and systemic conditions. PCOS, a hormonal disorder in women of reproductive age, often associates with obesity, dyslipidemia, and insulin resistance, heightening the risk for type 2 diabetes (T2D) and cardiovascular disease (CVD). The pathogenesis of PCOS involves an inflammatory response marked by increased CRP, inflammatory cytokines, elevated blood leukocytes, adhesion molecule expression, and oxidative stress markers like myeloperoxidase (MPO).

Periodontal diseases, bacterial infections affecting gums, ligaments, cement, and bone, include gingivitis (gum inflammation) and periodontitis (irreversible tissue destruction). Evidence suggests a link between periodontitis and increased CVD risk, while such association with gingivitis is limited.

Potential mechanisms linking periodontal diseases and CVD involve cytokine release, oral bacteria toxin production, and direct bloodstream transfer. Recognition of lipopolysaccharide (LPS) and TNFα triggers innate immune cells via TLR4 and TNFR, activating NF-κB and JNK expression. JNK amplifies inflammatory responses, inducing proinflammatory genes, and TNFα, IL-1, IL-6, and IL-8 can invade endothelial layers, promoting adhesion molecule expression. Enhanced leukocyte ROS production, especially in periodontitis, contributes to endothelial dysfunction and heightened cardiovascular risk.

The activation of multiple inflammatory pathways likely links PCOS, periodontal disease, and increased cardiovascular risk. Thus, the researchers aim to investigate if the presence of periodontal diseases, particularly gingivitis, exacerbates oxidative stress, inflammation and atherosclerosis surrogate markers in women with PCOS, and explore the underlying molecular mechanisms.

DETAILED DESCRIPTION:
The population will be identified using the Rotterdam criteria, which will include the following characteristics: irregular ovulation (cycles longer than 35 days or less than 26 days); elevated levels of free testosterone (>0.5 ng/dl; the cut-off level for free testosterone will be determined based on the mean ± 2 standard deviations from normal levels observed in the control group); hirsutism (total Ferriman-Gallwey score > 7); and the presence of polycystic ovaries, which will be identified through transvaginal ultrasonography (i.e., the presence of 12 or more small follicles measuring 2 to 9 mm in each ovary). The control group will be matched in BMI and age to the intervention group. In both groups, all medication, pathologies, and other medical conditions that could affect their reproductive physiology will be registered. All patients will receive detailed information on the study, highlighting its benefits and drawbacks, and will sign the informed consent and confidentiality commitment.

A comprehensive periodontal examination will be conducted across all study cohorts, adhering to established consensus criteria. Each tooth in the oral cavity will be probed at 6 points-3 buccal and 3 palatal-utilizing a periodontal chart with a Williams-type millimeter probe. Factors such as tobacco use, tooth brushing frequency, and alcohol consumption will be considered via a questionnaire, as well as through plaque and calculus indices. The periodontal examination will be carried out by a single doctor with training in periodontics to avoid inter-explorer bias. The researchers will also ask about dental treatments received, emphasizing periodontal treatments or those related to generating changes in soft tissues such as orthodontic gingival recessions. The periodontal measures will include the percentage of bleeding on probing (BOP), millimeters of clinical attachment level (CAL), millimeters of probing pockets depth (PPD), percentage of loss of bone, number of teeth with periodontal pockets-PPD ≥4mm- and number of teeth with CAL≥4mm-. The researchers will evaluate the plaque and calculus level using the Silness and Löe index for plaque and O´Leary index for calculus levels. To facilitate the measurement of plaque and calculus indexes, as they will be carried out in a hospital with a high flux of patients, these indices will be measured on the Ramfjord index teeth (right permanent maxillary first molar, right permanent incisor, left permanent first premolar, left mandibular permanent first molar, right permanent mandibular incisor, and right permanent mandibular first premolar).

A peripheral venous blood sample will be taken after 12 hours of fasting, during the follicular phase of the menstrual period of the patients (from the 1st to the 5th day of bleeding) to avoid biases dependent on the variability of sexual hormones. Neutrophils and PBMC will be isolated from 8 mL of EDTA-anticoagulated peripheral blood by means of an immunomagnetic method, following the manufacturer's protocol. In addition, LUNA-FL will be used to determine cell count and viability (acridine orange and propidium iodide double stain). Proteins will be extracted from neutrophils or PBMC on ice. Neutrophils will be lysed for 15 minutes with RIPA Lysis Buffer supplemented with protease and phosphatase inhibitors. The supernatant will be collected after centrifugation for 15 minutes at 16,000g. The total protein concentration will be quantified using a bicinchoninic acid (BCA) protein assay. Aliquots of 25µg of protein will be resolved on 8-16% gradient SDS-polyacrylamide gels and transferred to nitrocellulose membranes. Target proteins will be detected by incubating the membranes with anti-actin, JNK, NFkB, MCP1, GPX-1, NLRP3, ASC, procaspase 1, caspase 1, Beclin, ATG5-ATG12, p62, LC3 I, LC3 II, Pink1, GRP78, eIF2alpha, IRE1 alpha, ATF6, CHOP, PGC1 alpha, mTFA, VDAC, Complex I, II, III, IV and V. The protein signal will be detected by chemiluminescence and analyzed by densitometry.

A parallel plate flow chamber, connected to an inverted microscope, will enable the researchers to measure neutrophil-endothelial cell interactions in vitro. Prior to this, immortalized endothelial cells from the human umbilical vein will be seeded. One million leukocytes in 1 mL of RPMI medium will be drawn across the HUVEC. A video camera connected to the microscope will permit a 5 × 25 mm view of the endothelial cells. Various leukocyte parameters, including rolling velocity, rolling flux, and adhesion, will be evaluated over a period of 5 minutes. Analysis of serum cytokines, cellular adhesion molecules, and glutathione will be measured with a Luminex® 200 analyzer system following the Milliplex® MAP Kit manufacturer's procedure or ELISA technique.

This study was designed to achieve a power of 80% and to detect significant differences of 20 % in relation to the primary efficacy criterion - leukocyte-endothelium interactions (measured by adhesion of neutrophils) - assuming that 3 groups existed. Under these premises, at least 12 subjects per group were considered. Normally and non-normally distributed data will be expressed as mean ± standard deviation (SD) and median (25th-75th percentiles), respectively. Qualitative data will be expressed as percentages. The data will be analyzed using an unpaired Student's t test or a Mann-Whitney U test for parametric and non-parametric data, respectively. When comparing three groups, statistical significance will be assessed by one-way ANOVA or the Kruskal Wallis test followed by post hoc test. The strength of the association between variables will be measured by means of Pearson's or Spearman correlation coefficient, for parametric and non-parametric data, respectively. To predict the value of a variable based on another variable, linear regression analysis will be used. Differences will be considered significant when p < 0.05, with a confidence interval of 95%. Analysis will be performed with SPSS 22.0.

ELIGIBILITY:
Inclusion Criteria:

* Women with polycystic ovary syndrome (PCOS) according to the Rotterdam criteria:

  1. Irregular ovulation (cycles longer than 35 days or less than 26 days)
  2. Elevated levels of free testosterone (>0.5 ng/dl)
  3. Hirsutism and the presence of polycystic ovaries
* Healthy women without periodontal diseases matched in BMI and age to the PCOS group.

Exclusion Criteria:

* Other systemic inflammatory conditions
* Recent antibiotic use
* Chronic anti-inflammatory use
* Cancerous or bone-affecting pathologies
* Diabetes or autoimmune diseases
* Use of any medication during the previous semester

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — According to presence of polycystic ovary syndrome
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Evaluate subclinical atherosclerotic markers in the study population | At recruitment
  Determine leukocyte-endothelial cell interactions and cellular adhesion molecules in serum (ICAM, VCAM and p-Selectin)
Evaluate inflammatory markers in the study population | At recruitment
  Determine proinflammatory cytokines in serum (TNF-alpha, IL6) and expression of inflammatory mediators in leukocytes by Western blot (JNK, NFkB, MCP1)
Evaluate oxidative stress markers in the study population | At recruitment
  Determine serum oxidative stress markers (MPO, glutathione), expression of GPX-1 by Western blot and total ROS, mitochondrial ROS and superoxide by flow cytometry in leukocytes.

SECONDARY OUTCOMES:
Evaluate inflammasome complex activation in the study population | At recruitment
  Determine expression of NLRP3, ASC, procaspase 1 and caspase 1 by Western blot in leukocytes and serum levels of IL1 beta and IL18 in serum.
Evaluate markers of autophagy in the study population | At recruitment
  Determine expression of Beclin, ATG5-ATG12, p62, LC3 I, LC3 II and Pink by Western blot in leukocytes.
Evaluate markers of ER stress in the study population | At recruitment
  Determine expression of GRP78, eIF2alpha, IRE1 alpha, ATF6 and CHOP by Western blot in leukocytes.
Evaluate markers of mitochondrial biogenesis and complexes in the study population | At recruitment
  Determine expression of PGC1 alpha, mTFA, VDAC, Complex I, II, III, IV and V by Western blot in leukocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Milagros Rocha, PhD, Principal Investigator — FISABIO-HOSPITAL DR PESET
Locations (1):
- Hospital Universitario Doctor Peset, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marquez-Arrico CF, Silvestre-Rangil J, Gutierrez-Castillo L, Martinez-Herrera M, Silvestre FJ, Rocha M. Association between Periodontal Diseases and Polycystic Ovary Syndrome: A Systematic Review. J Clin Med. 2020 May 23;9(5):1586. doi: 10.3390/jcm9051586. PMID 32456146
- [Background] Romandini M, Baima G, Antonoglou G, Bueno J, Figuero E, Sanz M. Periodontitis, Edentulism, and Risk of Mortality: A Systematic Review with Meta-analyses. J Dent Res. 2021 Jan;100(1):37-49. doi: 10.1177/0022034520952401. Epub 2020 Aug 31. PMID 32866427
- [Background] Porwal S, Tewari S, Sharma RK, Singhal SR, Narula SC. Periodontal status and high-sensitivity C-reactive protein levels in polycystic ovary syndrome with and without medical treatment. J Periodontol. 2014 Oct;85(10):1380-9. doi: 10.1902/jop.2014.130756. Epub 2014 Mar 4. PMID 24592911
- [Background] Schenkein HA, Loos BG. Inflammatory mechanisms linking periodontal diseases to cardiovascular diseases. J Clin Periodontol. 2013 Apr;40 Suppl 14(0 14):S51-69. doi: 10.1111/jcpe.12060. PMID 23627334
- [Background] Greabu M, Giampieri F, Imre MM, Mohora M, Totan A, Pituru SM, Ionescu E. Autophagy, One of the Main Steps in Periodontitis Pathogenesis and Evolution. Molecules. 2020 Sep 22;25(18):4338. doi: 10.3390/molecules25184338. PMID 32971808
- [Background] Domon H, Takahashi N, Honda T, Nakajima T, Tabeta K, Abiko Y, Yamazaki K. Up-regulation of the endoplasmic reticulum stress-response in periodontal disease. Clin Chim Acta. 2009 Mar;401(1-2):134-40. doi: 10.1016/j.cca.2008.12.007. Epub 2008 Dec 13. PMID 19109937
- [Background] Paladines N, Dawson S, Ryan W, Serrano-Lopez R, Messer R, Huo Y, Cutler CW, Ramos-Junior ES, Morandini AC. Metabolic reprogramming through mitochondrial biogenesis drives adenosine anti-inflammatory effects: new mechanism controlling gingival fibroblast hyper-inflammatory state. Front Immunol. 2023 Jun 7;14:1148216. doi: 10.3389/fimmu.2023.1148216. eCollection 2023. PMID 37350964